CLINICAL TRIAL: NCT00790088
Title: International Report on Routine Practice of Sensor-enabled Pump Therapy
Brief Title: INTERPRET - International Report on Routine Practice of Sensor-enabled Pump Therapy
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: EUR04
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; continuous glucose monitoring; sensor-augmented pump therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — capillary blood samples for HbA1c analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the project is to document the international routine practice in sensor usage in patients treated with sensor-augmented pump therapy and to assess which variables (e.g. training of patients, frequency of sensor usage etc) are associated with an improvement in clinical outcome(s) from the start of the sensor use to the end of the follow-up period.

DETAILED DESCRIPTION:
Pump therapy has been established as "gold standard" for insulin delivery offering improvements over multiple daily insulin injections, but there is a proportion of patients for whom the Continuous Subcutaneous Insulin Infusion (CSII) has not been completely successful therapy leaving some room for improvement of the glucose level of those patients. Continuous glucose monitoring (CGM) systems represent an important advance in diabetes technology that can facilitate optimal glucose control in type 1 diabetes. Numerous randomized control trials have demonstrated the safety and efficacy of real-time CGM in both sub-optimally and well-controlled type 1 diabetes. In all these trials, the benefits of CGM correlate with frequent sensor wear and more advanced age. In clinical practice, the sensor-augmented pump therapy (SAP therapy) is indicated for patients who cannot achieve good metabolic control on CSII, who have a history of severe hypoglycemia and/or hypoglycemia unawareness, or who desire increased flexibility in their daily lives while maintaining or even improving their HbA1c levels.

This was a post-market release, minimally interventional study. All the study devices and related software were CE-marked and commercially available in the countries participating to the study. The devices were prescribed and reimbursed, if applicable, according to routine practice.

The gathered information during this study may help to define which patient groups benefit the most from the treatment with SAP therapy systems. The real-life results of these descriptive analyses will aid improvement of guidelines helping the medical community to better choose the right patient population and treatment patterns. Moreover, based on these real-life data, hypotheses could be defined when addressing further research questions.

ELIGIBILITY:
Inclusion Criteria:

* Patient (and/or legal representative) has signed Patient Informed Consent (PIC)
* Patient was diagnosed with Type 1 DM and has been on insulin infusion pump therapy (without any additional insulin injection) for at least 6 months prior to signature of the PIC
* The treating physician decided independently of the study to prescribe non-blinded continuous glucose monitoring as part of the patient's pump therapy for at least 10% of the study time (estimated as days per month)

Exclusion Criteria:

* Participation in any other clinical trial - currently and/or in the last 3 months prior to signature of informed consent
* Patient has preliminary experience with non-blinded continuous glucose monitoring prior to signature of informed consent (not naïve to non-blinded continuous glucose monitoring)
* For children: no reliable contact person

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 diabetes on insulin infusion pump therapy
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Cohen, Prof, Principal Investigator — Chaim Sheba Medical Center, Tel Hashomer, Israel; Kirsten Noergaard, MD, Principal Investigator — Hvidovre Hospital, Hvidovre, Denmark; Andrea Scaramuzza, MD, Principal Investigator — Sacco Hospital, University of Milan, Italy
Locations (26):
- LKH Salzburg/Universitätsklinikum der Paracelsus Med Privatuniversität/Innere Medizin I, Salzburg, Austria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - AZ Imelda, Bonheiden
- Denmark (2):
  - Fredericia Hospital, Fredericia
  - Hvidovre Hospital, Hvidovre
- France (3):
  - Hôpital de Dax, Dax
  - Centre Hospitalier de Haguenau, Haguenau
  - Centre Hospitalier La Rochelle, La Rochelle
- Hungary (3):
  - Réthy Pál Hospital, Békéscsaba
  - Péterfy Hospital, Outpatient Clinic, Budapest
  - Josa András Teaching Hospital, Nyíregyháza
- Chaim Sheba Medical center, Tel Hashomer, Ramat Gan, Israel
- Italy (2):
  - Sacco Hospital, University of Milan, Milan
  - Ospedale S. Camillo Forlanini, Roma
- Kaunas University Hospital, Kaunas, Lithuania
- Poland (3):
  - Klinika Chorób Dzieci Uniwersytecki Dzieciecy Szp, Bialystok
  - Specjalistyczna Praktyka Lekarska, Gliwice
  - Oddzial Kliniczny Kliniki Chorób Metabolicznych Sz, Krakow
- Clinical Center of Serbia, Belgrade, Serbia
- Slovakia (2):
  - TopCare s.r.o., Košice
  - National Institute of Endocrinology, Ľubochňa
- University Childrens Hospital, Ljubjana, Slovenia
- Spain (3):
  - Hospital Universitario Infanta Cristina, Badajoz
  - Complejo Hosp. Santiago De Compostela, Santiago de Compostela
  - Hospital Virgen del Rocio, Seville
- Astrid Lindgrens Barnsjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Nørgaard K et al. Routine sensor-augmented pump therapy in type 1 diabetes: the INTERPRET study. Diabetes Technol Ther. 2013 Apr;15(4):273-80. doi: 10.1089/dia.2012.0288. Epub 2013 Feb 25.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At baseline, few patients had to be excluded from analyses due to major protocol deviations such as missing patient informed consent, CSII therapy for less than 6 months, prior experience with SAP therapy, and no eCRF data information available. Hence 263 patients were eligible for analyses at baseline.
Groups:
- Sensor-augmented Pump: CSII patient who were prescribed the use of continuous glucose monitoring (CGM) for at least 10% of the time
Period: Overall Study
Arm/Group | Sensor-augmented Pump
Started | 274
Eligible for Data Analysis | 263 (Number of participants minus 11 protocol violation)
Completed | 235
Not Completed | 39
Not completed — Protocol Violation | 11
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sensor-augmented Pump
Number analyzed (Participants) | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.04 (15.72)
Age, Customized [Number; unit: participants] — Age groups are: 0-7; 8-12; 13-17; 18-24; >24
  participants
    <=7 years | 28
    8 - 12 | 21
    13-17 | 35
    18-24 | 27
    >24 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 99
Region of Enrollment [Number; unit: participants]
  Serbia | 20
  Slovenia | 20
  Spain | 22
  Lithuania | 14
  Austria | 4
  Israel | 14
  Italy | 18
  Slovakia | 4
  France | 22
  Poland | 39
  Hungary | 17
  Belgium | 20
  Denmark | 28
  Sweden | 12
  Czechia | 9

OUTCOME MEASURES:

1. Primary Outcome: Frequency as Percentage of Sensor Usage
Description: To calculate the percentage of time that sensors were used during 3 months:
  the total number of recorded sensor readings during 3 months was divided by the theoretical number of sensor readings that would be observed if sensor was worn every day of using pump to deliver insulin during the same period (ie, observed readings / (theoretical 288 readings per day x nber of days with insulin use)) and multiplied by 100
Time Frame: every 3 months
Measure: Mean (Standard Deviation); unit: % of time
Groups:
- Whole Population: all available data from eligible patients at baseline
Arm/Group | Whole Population
Number analyzed (Participants) | 263
% of time
  Baseline - 3 months | 37 (29)
  3 months - 6 months | 31 (28)
  6 months - 9 months | 28 (28)
  9 months - 12 months | 27 (28)
  baseline - 12 months | 30 (26)

2. Primary Outcome: HbA1c
Time Frame: every 3 months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Sensor-augmented Pump
Number analyzed (Participants) | 263
percent
  Baseline | 8.1 (1.4)
  3Months | 7.87 (1.2)
  6Months | 7.9 (1.17)
  9Months | 7.98 (1.14)
  12Months | 8.05 (1.23)

3. Primary Outcome: Percentage of Patients Achieving HbA1c < 7%
Time Frame: every 3 months
Measure: Number; unit: percent of patients
Arm/Group | Sensor-augmented Pump
Number analyzed (Participants) | 263
percent of patients
  Baseline | 18.25
  3 months | 18.5
  6 months | 18.22
  9 months | 17.72
  12 months | 16.02

4. Secondary Outcome: Fear of Hypoglycemia Survey (HFS-II) - Total Score and Behavior Score
Description: sub-group of patients (adults only in Hungary and Denmark) were asked to answer the fear of hypoglycemia validated questionnaires.
  The total HFS-II questionnaire is represented by 33 items. The respondents rank the responses on a 5- point Likert scale where zero is never and four is always.The total HFS-II score ranges from 0 to 132. Lower score at 6 months or 12 months compared to baseline represents a better outcome.
  The HFS-II questionnaire is divided into 2 subscales: the behavior and the worry subscales. The behavior score is represented by 15 items and ranges from 0 to 60. Lower score at 6 months or 12 months compared to baseline represents a better outcome.
Time Frame: at baseline, after 6 and after 12 months
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Whole Population
Number analyzed (Participants) | 40
Score
  Total score at baseline | 37 (25.94)
  Total score at 6Months | 32.74 (21.24)
  Total score at 12Months | 28.95 (20.11)
  Behavior Score at baseline | 16.03 (10.71)
  Behavior score at 6Months | 14.56 (9.06)
  Behavior score at 12Months | 13.35 (8.81)

5. Secondary Outcome: Fear of Hypoglycemia Survey (HFS-II) - Worry Score
Description: sub-group of patients (adults only) were asked to answer the fear of hypoglycemia validated questionnaires. The respondents rank the responses on a 5- point Likert scale where zero is never and four is always. The worry subscale is the mean of 18 items which evaluate the worry score (range from 0 to 72). Lower score at 6 months or 12 months compared to baseline represents a better outcome.
Time Frame: at baseline, after 6 and after 12 months
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Whole Population
Number analyzed (Participants) | 61
Score
  Worry score at baseline | 23.39 (15.65)
  Worry score at 6Months | 20.65 (15.37)
  Worry score at 12Months | 18.40 (14.84)

6. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire Status Version (DTSQs)
Description: A sub-group of patients (adults) were asked to complete the Diabetes Treatment Satisfaction Questionnaire (DTSQs) The treatment satisfaction is measured by means of the Diabetes Treatment Satisfaction Questionnaire, status version (DTSQs, Bradley, 1990). It consists of a six-item scale assessing treatment satisfaction (TS) and two items assessing perceived frequency of hyperglycaemia and hypoglycaemia. The DTSQs items are scored on a scale from 6 to 0. The scale total is computed by adding the six items 1, 4, 5, 6, 7, and 8, to produce the Treatment Satisfaction scale total, which has a min of 0 and a max of 36. Higher score at 6 month or 12 months compared to baseline represents a better outcome. Items 2 (perceived frequency of hyperglycaemia) and 3 (perceived frequency of hypoglycaemia) are treated individually in data analysis. Lower score at 6 months or 12 months compared to baseline represents a better outcome.
Time Frame: at baseline, after 3 and after 12 months
Measure: Mean (Standard Deviation); unit: score
Groups:
- SAP Users: Patients in Spain, Denmark and Hungary participated, where the questionnaires translations were validated
Arm/Group | SAP Users
Number analyzed (Participants) | 66
score
  Diatbetes Treatment satisfaction score at baseline | 31.42 (3.15)
  Treatment satisfaction score at 3Months | 30.80 (4.33)
  Treatment satisafaction score at 12Months | 32 (3.29)
  Perceived Frequency Hypoglycaemia at baseline | 2.18 (1.28)
  Perceived Frequency Hypoglycaemia at 3Months | 2.5 (1.32)
  Perceived Frequency Hypoglycaemia at 12Months | 2.03 (1.16)
  Perceived Frequency Hyperglycaemia at baseline | 2.83 (1.30)
  Perceived Frequency Hyperglycaemia at 3Months | 2.67 (1.17)
  Perceived Frequency Hyperglycaemia at 12Months | 2.35 (1.33)

7. Primary Outcome: Percentage of Patients Achieving HbA1c < 7.5%
Time Frame: every 3 months
Measure: Number; unit: percent of patients
Arm/Group | Sensor-augmented Pump
Number analyzed (Participants) | 263
percent of patients
  Baseline | 28.52
  3 months | 36.22
  6 months | 32.79
  9 months | 31.65
  12 months | 33.33

ADVERSE EVENTS:
Time Frame: During the 12Months follow-up
Description: Only Serious adverse events were collected
Arm/Group | Sensor-augmented Pump
Serious Adverse Events (participants affected / at risk) | 24/263
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor-augmented Pump (N=263)
Diabetic ketoacidosis (Endocrine disorders) | 3 (3) — defined as blood glucose >250 mg/dL [>13.9 mmol/L] with either low serum bicarbonate [<15 mEq/L] or low pH [<7.3] and either ketonemia or ketonuria and requiring treatment within a health-care facility
Severe hypoglycemia (Endocrine disorders) | 9 (13) — defined as an episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory blood glucose value <50mg/dL [<2.8 mmol/L]
Other diabetes-related AE (Endocrine disorders) | 6 (6) — angioplasty, diabetic foot ulcer; ischemic heart disease; pancreas and liver transplantations, suicide attempt, poor glycemic control
Non Diabetes-related serious adverse events (Endocrine disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less